CLINICAL TRIAL: NCT00721071
Title: Diagnostic Utility of Induced Sputum Using Hypertonic Saline to Evaluate Airway Infection and Inflammation in Cystic Fibrosis
Brief Title: Utility of Induced Sputum Using Hypertonic Saline to Evaluate Infection and Inflammation in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000009154
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cystic Fibrosis
Keywords: Pediatrics; Cystic Fibrosis; Hypertonic Saline; Induced Sputum; Expectorated Sputum
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Hypertonic Saline

INTERVENTIONS:
Drug: Hypertonic Saline — After each subject has performed post-bronchodilator spirometry, he/she will inhale increasing concentrations of 3, 4, and 5% of hypertonic saline for 7 minutes each for 3 cycles until expectorating a sufficient sputum sample.

SUMMARY:
The objective of the study is to evaluate the clinical utility and the feasibility, in an outpatient setting, of sputum induction using hypertonic saline. This study will also study pilot techniques on a sub using a sub-sample to assess the lower airway inflammatory cells and markers in relation to new emerging organisms in cystic fibrosis (CF) and antibiotic therapy in CF.

DETAILED DESCRIPTION:
Chronic airway infection, mainly by Staphylococcus aureus (SA) and Pseudomonas aeruginosa (PA), is a major cause of morbidity and mortality in patients with cystic fibrosis (CF). Isolation of organisms from the respiratory tract is important to optimize treatment. The current recommended methods for bacterial evaluation are bronchoalveolar lavage (BAL) and expectorated sputum (ES) analysis. However, a significant proportion of young CF patients cannot produce sputum spontaneously. The method used most frequently therefore is to isolate respiratory organisms is to perform throat swabs (TS) which have poor sensitivity and specificity in the evaluation of respiratory pathogens in CF patients.

Induced sputum (IS) using hypertonic saline has been used in a limited number of studies to evaluate respiratory organisms in CF patients. These studies have reported that IS may be a useful non-invasive diagnostic test to increase the yield of detection of respiratory pathogens.

Beside its use as a diagnostic test to identify bacterial pathogens induced sputum has been used to assess lower airway inflammation in CF. While numerous studies have clarified the role of S. aureus and P. aeruginosa in CF lung disease, the role of other emerging bacteria such as Stenotrophomonas maltophilia (SM) and Achromobacter xylosoxidans (AX) species remains largely unclear. IS offers the potential to possibly differentiate between colonisation and infection for the emerging pathogens and to help clarify their role in CF lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with CF (by sweat chloride ≥60 and/or genetic testing)
2. Children ages between 6-18 years
3. Ability to perform pulmonary function tests
4. FEV1 ≥ 30% predicted18.

Additional inclusion criteria for sub-sample undergoing antibiotic therapy:

1. Above criteria
2. Admitted to hospital for i.v. antibiotic therapy

Exclusion Criteria:

1. Acute respiratory distress or hypoxia (oxygen saturation <92% at room air)
2. New onset of wheezing
3. Previous history of intolerance of inhalation of HS

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Additional positive bacterial culture yield post IS technique for known and emerging CF pathogens over conventional methods of bacterial culturing (ES and TS). | 60 minutes; for subgroup, this will be repeated a second time after 14 days.

SECONDARY OUTCOMES:
Inflammatory profile as measured by relative neutrophil count and IL-8 concentration in the IS | 60 minutes; for subgroup, this will be repeated a second time after 14 days.
Bacterial colony counts | 60 minutes; for subgroup, this will be repeated a second time after 14 days.
Frequency of change in clinical management based on results from IS | 60 minutes; for subgroup, this will be repeated a second time after 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Al-Saleh S, Dell SD, Grasemann H, Yau YC, Waters V, Martin S, Ratjen F. Sputum induction in routine clinical care of children with cystic fibrosis. J Pediatr. 2010 Dec;157(6):1006-1011.e1. doi: 10.1016/j.jpeds.2010.06.001. Epub 2010 Jul 14. PMID 20630539